CLINICAL TRIAL: NCT03544138
Title: Pivotal Study of the Preceptis Medical Inc. Hummingbird™ Tympanostomy Tube System (H-TTS) in the Otolaryngology Clinic
Brief Title: In-Office Study of the Hummingbird® in Children 6 Months-21 Years Old
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Preceptis Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Preceptis Pivotal
Record Dates: First submitted 2018-05-09; First posted 2018-06-01 (Actual); Results first posted 2022-12-14 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-11

CONDITIONS: Ear Infection; Otitis Media
MeSH Terms: conditions — Otitis; Otitis Media

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Hummingbird Tympanostomy Tube System (H-TTS) (Other): The Hummingbird Tympanostomy Tube System (H-TTS) is a disposable surgical tool designed to deliver a tympanostomy tube ("ear tube") into the tympanic membrane of patients during a tympanostomy tube placement procedure.
  Interventions: Device: Hummingbird Tympanostomy Tube System (H-TTS)

INTERVENTIONS:
Device: Hummingbird Tympanostomy Tube System (H-TTS) — The H-TTS is intended to deliver a tympanostomy tube through the tympanic membrane of a patient during a tympanostomy procedure.
  Other Names: H-TTS

SUMMARY:
The objective of this study is to evaluate the safety and performance of the Hummingbird® for the placement of ear tubes in children undergoing tympanostomy tube placement in an otolaryngology clinic using local anesthetic.

DETAILED DESCRIPTION:
The Hummingbird Tympanostomy Tube System (H-TTS) is intended to deliver a tympanostomy tube (also referred to as a ventilation tube) through the tympanic membrane of the patient and is indicated to be used in office settings for children. The H-TTS is intended to deliver a tympanostomy tube through the tympanic membrane (TM) of the patient. It combines the separate functions of creating a myringotomy, and positioning and placing a ventilation tube across the TM.

The Hummingbird Tympanostomy Tube System (H-TTS) is a disposable surgical tool designed to deliver a tympanostomy tube ("ear tube") into the tympanic membrane of patients during a tympanostomy tube placement procedure. More than 1,000,000 ear tubes are inserted annually in the US, making it one of the most common surgical procedures performed in children.

Preceptis Medical, Inc. has developed the H-TTS to reduce trauma, pain, and risk to the patient while reducing the overall surgical procedure time. The H-TTS integrates the multiple surgical instruments necessary for current surgical procedure into a single, one-pass device. The H-TTS creates an incision in the tympanic membrane ("ear drum") and inserts a tympanostomy tube with the push of a lever. Thus, the H-TTS allows placement of a tympanostomy tube with a single pass down the ear canal. The ear tube used with the H-TTS is a standard, commercially available tympanostomy tube.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo tympanostomy tube insertion in the clinic.
* Children 6 months to 21 years old
* Signed parental consent, and child assent documents as applicable.
* Parent is fluent in English.

Exclusion Criteria:

* Any condition that, in the opinion of the investigator, may place the subject at greater risk (e.g., child with developmental delay).
* Anatomy precludes sufficient visualization and access to the tympanic membrane.

Ages: 6 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 258 (Actual)
Dates: Start 2018-07-24 (Actual); Primary Completion 2022-09-06 (Actual); Study Completion 2022-09-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Cedars-Sinai Medical Care Foundation, Beverly Hills, California
  - Children's Ear Nose Throat & Allergy, Orlando, Florida
  - HealthPartners Institute, Bloomington, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - St. Cloud Ear, Nose & Throat, Saint Cloud, Minnesota
  - Park Nicollet, Saint Louis Park, Minnesota
  - Prairie Sinus Ear & Allergy, P.C., Bismarck, North Dakota

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available to other researchers.

REFERENCES:
- [Derived] Truitt TO, Kosko JR, Nimmons GL, Raisen J, Skovlund SM, Rimell F, Cofer SA. In-office insertion tympanostomy tubes in children using single-pass device. Laryngoscope Investig Otolaryngol. 2021 Feb 2;6(2):325-331. doi: 10.1002/lio2.533. eCollection 2021 Apr. PMID 33869765
- See also: Precepts Medical, Inc. — https://www.preceptismedical.com

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Number of ears
Groups:
- Hummingbird Tympanostomy Tube System (H-TTS) Tube Delivery: Subjects will have ear tubes placed with the Hummingbird Tympanostomy Tube System (H-TTS) in an office setting using topical anesthetic.
Period: Overall Study
Arm/Group | Hummingbird Tympanostomy Tube System (H-TTS) Tube Delivery
Started | 258; 492 Number of ears (Number of participants and ears that underwent ear tube placement with HTTS.)
Completed | 229; 440 Number of ears (Number of participants and ears that completed follow-up at 3-10 weeks post-procedure)
Not Completed | 29; 52 Number of ears
Not completed — Lost to Follow-up | 29

BASELINE CHARACTERISTICS:
Arm/Group | Hummingbird Tympanostomy Tube System (H-TTS)
Number analyzed (Participants) | 258
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 258
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110
  Male | 148
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 258

OUTCOME MEASURES:

1. Primary Outcome: Rate of Ears Experiencing an Adverse Events From Enrollment to 3-10 Week Follow-up
Description: AEs that occurred from enrollment through the 3-10 week follow-up were collected.
Time Frame: Follow-up between 3-10 weeks
Population: Rate of ears experiencing an adverse event. There were 258 participants and 492 ears analyzed.
Measure: Number; unit: percentage of ears
Units Other Than Participants: Ears
Arm/Group | Hummingbird Tympanostomy Tube System (H-TTS)
Number analyzed (Participants) | 258
Number analyzed (Ears) | 492
percentage of ears | 0.41

2. Primary Outcome: Percentage of Ears With Successful Delivery of the Tympanostomy Tube by the H-TTS
Description: Efficacy evaluation will consist of determining whether the H-TTS device successfully delivers the tympanostomy tube across the tympanic membrane.
Time Frame: Intra-Procedure
Measure: Number; unit: percentage of ears
Units Other Than Participants: Ears
Arm/Group | Hummingbird Tympanostomy Tube System (H-TTS)
Number analyzed (Participants) | 258
Number analyzed (Ears) | 492
percentage of ears | 97.2

3. Primary Outcome: Percentage of Participants With Successful Completion of Procedure In-office
Description: Success will be defined as the ability of the surgeon to place ear tubes using the H-TTS device in the office setting with the use of local anesthetic.
Time Frame: Intra-procedure
Measure: Number; unit: percentage of participants
Arm/Group | Hummingbird Tympanostomy Tube System (H-TTS)
Number analyzed (Participants) | 258
percentage of participants | 98.4

ADVERSE EVENTS:
Time Frame: All adverse events (AE), both anticipated and unanticipated, were reported through follow-up of 3-10 weeks.
Arm/Group | Hummingbird Tympanostomy Tube System (H-TTS)
All-Cause Mortality (participants affected / at risk) | 0/258
Serious Adverse Events (participants affected / at risk) | 0/258
Other Adverse Events (participants affected / at risk) | 1/258
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hummingbird Tympanostomy Tube System (H-TTS) (N=258)
Acute tube extrusion (Surgical and medical procedures) | 1 (1) — During the surgical procedure, a myringotomy incision is completed but the tympanostomy tube will not stay in the tympanic membrane.
Tube dislocating into middle ear space (Surgical and medical procedures) | 1 (1) — Tube passes completely through the tympanic membrane and falls into the middle ear cavity and is unable to be retrieved in office

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-29): https://cdn.clinicaltrials.gov/large-docs/38/NCT03544138/Prot_SAP_000.pdf